CLINICAL TRIAL: NCT04734444
Title: Ultrasound Imaging in Brain Tumour Surgery With the Use of SonoClear Acoustic Coupling Fluid (ACF) Mimicking Brain Tissue
Brief Title: SonoClear Acoustic Coupling Fluid (ACF) Mimicking Brain Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SonoClear AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACF-03
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumour; High Grade Glioma; Low-grade Glioma; Glioblastoma
Keywords: Acoustic Coupling Fluid (ACF); Ultrasound imaging in brain tumour surgery; brain tumour surgery
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma

STUDY DESIGN:
Intervention Model Description: A prospective, multi-centre single arm study
Masking Description: The following measures have been taken to minimize or avoid bias:
  * Core-lab evaluation of the CNR outcome in a blinded fashion
  * SIR clinical rating of US images by an independent expert panel in a blinded fashion
  Due to the nature of brain surgery and the diversity of the tumours, it is seen as a strength to the trial that the patient can act as its own control even though the images can never be 100% the same in the separate image acquisition. This is especially true for 2D US images, whereas with a 3D US image it is more likely to obtain the same position for sequential image acquisition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SonoClear acoustic coupling fluid (ACF) mimicking brain tissue (Experimental): SonoClear
  Interventions: Device: SonoClear ACF

INTERVENTIONS:
Device: SonoClear ACF — The SonoClear ACF is intended to be used as an acoustic coupling fluid during ultrasound imaging in brain surgery of human beings

SUMMARY:
The objective of this clinical investigation is to assess the safety and performance of the SonoClear Acoustic Coupling Fluid (ACF). The performance will be assessed by analysis of the contrast-to-noise ratio (CNR) and assessment of image quality by using the Surgeon Image Rating (SIR) Scale.

This is a prospective, multi-centre single-arm study where the performance of SonoClear ACF relative to routinely used acoustic coupling fluid is investigated by each patient being their own control. Patients with the diagnosis of HGG and LGG at up to 10 sites will be included. Additionally, safety data are collected at 30 days and 6 months post-procedure.

DETAILED DESCRIPTION:
Ultrasound images will be obtained at different timepoints during the operation. First timepoint being after craniotomy (no fluids involved). Second timepoint being when some tumour is left in the bottom of the deeper part of the resection cavity (approximately 80% of tumour removed), and third timepoint being when the surgeon deems resection of the tumour to be completed. At the second and third timepoint ultrasound acquisition will be performed twice at each timepoint. Once with routinely used saline / Ringer's solution and once with SonoClear ACF.

There are two performance related primary endpoints, based on core lab assessments:

1. To show that ultrasound images obtained with SonoClear ACF are less influenced by image artefacts compared to images obtained with standard of care saline or Ringer´s solution, by measuring the contrast-to-noise ratio (CNR). The CNR is a measure of the relative noise in the image. To achieve this endpoint, the use of SonoClear ACF must lead to superior image quality in comparison with Saline/Ringer´s solution. Superior image quality is defined as the CNR being statistically different between the images obtained with saline/Ringer and SonoClear ACF respectively, i.e., significantly less noise in the images obtained with SonoClear ACF.
2. To show that ultrasound images obtained with SonoClear ACF are of better quality compared to images obtained with standard of care Saline/Ringer's solution, by using a qualitative assessment, called the Surgeons Image Rating (SIR) scale. A Panel of Experts will assess the quality of the obtained images by answering 3 questions for each image. The SIR a 1-10 numeric rating scale, is used to measure the quality of the image according to three questions to be answered at the three different timepoints during the operation.

This SIR is designed to explore whether SonoClear ACF, having shown to provide better quantitative image quality in the CNR analysis, allows surgeons to detect this improved image quality. Eventually this improved image quality should result in better decision-making during surgery about margins of excision and residual tumour resection.

Primary Safety Endpoint

The primary safety hypothesis is to prove the primary safety event rate is less than 10%. The primary safety event is defined as any core lab determined major MRI finding when post-operative MRI is compared to pre-operative MRI that was found by the DMC to be serious and probably or definitely related to the study device OR any DMC determined serious adverse event that is probably or definitely related to the study device that occurs within 30 days of the procedure. Success is demonstrated by observing 0 of these events out of 37 subjects exposed to SonoClear ACF. This is equivalent to a two-sided p-value less 0.05 for the alternative hypothesis that the primary safety event rate in subjects undergoing tumor resection using ACF is less than 10%.

ELIGIBILITY:
Inclusion Criteria:

* A diffuse malignant glial tumour (high (grade III and IV) or low grade (grade I-II) is suspected from the diagnostic MRI scan
* A tumour that extends at least 3 cm in depth from the surface of the brain (confirmed by MRI)
* Pre- or peri-procedural confirmed histopathology of glioma
* ≥18 years of age
* Karnofsky performance status ≥ 70
* Life expectancy of more than 30 days at the time of the procedure
* Negative pregnancy test for female subjects of childbearing potential

Exclusion Criteria:

* Not able to give consent (e.g. severe cognitive impairment)
* History of brain radiation therapy
* Recent meningitis (within 6 months prior to screening visit)
* Other active infection (within 30 days prior to screening visit)
* Immuno-incompetent patient (e.g. failing immune system due to AIDS)
* Patients taking immune-suppressive medication
* Intended biopsy only (meaning: cases not suitable for resection)
* Known hypersensitivity to egg protein
* Known hypersensitivity to soybean or peanut protein
* Known Hypersensitivity to glycerol
* Known Hypersensitivity to polysorbates
* Pregnant or lactating females or females who intend to become pregnant during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Contrast-to-Noise Ratio (CNR) to quantify the reduction in noise | During ultrasound guided brain tumour resection
  To show that ultrasound images obtained when using SonoClear ACF are less influenced by image artefacts compared to images obtained when using routinely used saline solution measuring the contrast-to-noise ratio (CNR) in the images.
Surgeons Image Rating (SIR) to assess the image quality | During ultrasound guided brain tumour resection
  Quality assessment of the images is done by the core-lab in a blinded manner using the Surgeon Image Rating (SIR) scale, a 1-10 rating scale to score the quality of the image according to 3 questions at different time points during the operation. First timepoint being after craniotomy (no fluids involved). The second time point is when some tumour is left in the bottom of the deeper part of the resection cavity (approximately 80% of tumour removed), and the third time point being when the surgeon deems resection of the tumour to be completed.
Adverse events up to 30 days post procedure | safety data are collected up to 30 days post procedure
  The primary safety hypothesis is to prove the primary safety event rate is less than 10%. A primary safety event is defined as any core lab determined major MRI finding when post-operative MRI is compared to pre-operative MRI that was found by the DMC to be serious and probably or definitely related to the study device OR any DMC determined serious adverse event that is probably or definitely related to the study device that occurs within 30 days of the procedure. Success is demonstrated by observing 0 of these events out of 37 subjects exposed to SonoClear ACF. This is equivalent to a two-sided p-value less 0.05 for the alternative hypothesis that the primary safety event rate in subjects undergoing tumor resection using ACF is less than 10%.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (2):
  - Universitätsklinikum Ulm, Günzburg
  - Philipps-Universität Marburg, Marburg
- Instituto Neurologico "C. Besta", Milan, Italy
- University Hospital Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No